CLINICAL TRIAL: NCT04099082
Title: Signature of the Host Response to a Respiratory Viral Infection, in the Prediction of Bronchiolitis Obliterans
Acronym: ALLOPIV
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180175
Record Dates: First submitted 2019-08-19; First posted 2019-09-23 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell Recipients; Acute Respiratory Infection; Parainfluenza Virus (PIV)
MeSH Terms: interventions — Sampling Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: eligible patients with 10% decline in Forced Expiratory Volume (FEV1) at 2 months
  Interventions: Other: samples
- Controls: eligible patients free of 10% FEV1 decline at 2 months
  Interventions: Other: samples

INTERVENTIONS:
Other: samples — blood sample nasal swab

SUMMARY:
Bronchiolitis obliterans (BO) is the well-known manifestation of the chronic pulmonary graft-versus-host disease(GVHD) after allogeneic hematopoietic stem cell transplantation (HSCT). The pathophysiology of BO is, however, poorly known. The available data strongly support the role of respiratory viruses, in particular paramyxoviruses (parainfluenzae virus (PIV), respiratory syncytial virus, metapneumovirus). It is likely that the alloimmune response triggered by the respiratory virus is inadequate and leads to the peribronchiolar fibrotic process. The objective is to analyze the kinetics of profiles of the blood and respiratory host responses resulting from a high or low parainfluenza respiratory infection, in order to evaluate if the occurrence of a BO is associated with a specific signature We will evaluate the predictive signature of a BO after a parainfluenza virus infection by characterizing the differences between the patients evolving and those not evolving to a BO at 2 months after the infection.

ELIGIBILITY:
Inclusion Criteria :

* Adults having received a hematopoietic stem cell transplantation for less than two years
* Availability of respiratory function tests prior to infection
* Presence of PIV respiratory infection documented by identification of the virus by PCR in the upper and/or lower respiratory tract
* Symptoms of respiratory infection ≤ 5 days
* Signed informed consent

Exclusion Criteria:

* Presence of a respiratory virus infection other than PIV
* Viral respiratory co-infections
* Bacterial or fungal respiratory infections
* Treatment with ribavirin, oseltamivir or any other antiviral with activity against respiratory viruses
* Patient not affiliated or beneficiary of a social security system
* Patient deprived of liberty or protected
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult recipients of allogeneic HSCT with PIV pulmonary infection
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Host response in both blood and respiratory tract after PIV infection | Up to 6 months

SECONDARY OUTCOMES:
Identify the cellular signaling pathways associated with the development of BO following parainfluenzae virus infection | Up to 6 months
Evaluate differences in transcriptomic profiles between blood and respiratory tract | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided